CLINICAL TRIAL: NCT03941574
Title: A Single-arm, Multi-center, Phase Ⅱ Clinical Study to Evaluate the HLX10 Monotherapy for the Treatment of Unresectable or Metastatic Microsatellite Instability-high (MSI-H) or Mismatch Repair Deficient (dMMR) Solid Tumors That Failed to Respond to Standard Therapy
Brief Title: A Clinical Study to Evaluate HLX10 Monotherapy for the Treatment of MSI-H or dMMR Solid Tumors That Failed to Respond to Standard Therapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HLX10-010-MSI201
Record Dates: First submitted 2019-04-24; First posted 2019-05-08 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: MSI-H Solid Malignant Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HLX10 (Experimental)
  Interventions: Drug: HLX10

INTERVENTIONS:
Drug: HLX10 — HLX10 developed by our company is sterile intravenous injection, with specification of 100 mg/10 mL/bottle. The main ingredient is 10.0 mg/mL of recombinant humanized anti-PD-1 monoclonal antibody. The excipients include 0.95 mg/mL citric acid (citric acid monohydrate), 4.56 mg/mL sodium citrate (sodium citrate dihydrate), 3.0 mg/mL sodium chloride, 30.0 mg/mL mannitol and 0.20 mg/mL polysorbate 80 (tween 80), with pH of 5.5.

SUMMARY:
It is a single-arm, open-label, multicenter, phase II clinical study to evaluate the clinical efficacy and safety of HLX10 monotherapy for the treatment of patients with unresectable or metastatic MSI-H or dMMR solid tumors who have progressed or intolerable after standard therapy.This study consists of three periods, screening period (28 days), treatment period and follow-up period (including safety follow-up, survival follow-up).Subjects can be enrolled into this study only if they meet inclusion criteria and do not meet exclusion criteria. The enrolled subjects will receive an intravenous infusion of HLX10 (3 mg/kg) once every 2 weeks until the loss of clinical benefit, death, intolerable toxicity, withdrawal of informed consent or other reasons as specified in the protocol, or up to the longest treatment duration-2 years (52 dosing periods) (whichever occurs earlier).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who meet all of the following criteria are allowed to be enrolled into this study:

  * Volunteer to participate in this clinical study; completely understand and know this study as well as sign the informed consent form (ICF); be willing to follow and be able to complete all study procedures;
  * Age ≥ 18 years and ≤ 75 years when ICF is signed;
  * Patients with unresectable or metastatic MSI-H or dMMR malignant solid tumors which are histopathologically or/and cytologically confirmed by the central laboratory or study sites;
  * Patients who have disease progression or intolerable reactions after the currently available standard anti-cancer treatment previously received;
  * The interval between the end of previous systemic anti-tumor treatment and the first dosing of if this study must be ≥ 2 weeks. In addition, treatment-related AEs recover to NCI-CTCAE v4.03 ≤ grade 1 (excluding grade 2 alopecia).
  * There is at least one measurable lesion assessed by IRRC according to the requirements of RECIST version 1.1 (Appendix 1).

Note: measurable lesions cannot be selected from the previous radiotherapy sites. If the target lesion of the previous radiotherapy sites is the only one available lesion, the investigator is required to provide imaging data before and after significant progression of such lesion.

• Subjects must provide tumor tissues and blood samples for the determination of MSI, tumor mutational burden (TMB), PD-L1 expression level (if the test results of the above parameters by the central laboratory specified by this study are available, the subjects are allowed not to receive repeated tests).

Note: it is recommended to provide formalin fixed tumor tissue samples collected from non-radiotherapy sites within 6 months prior to the first dosing of investigational product, paraffin embedded tumor samples (preferred), or formalin fixed paraffin embedded tumor samples or unstained newly sliced serial sections (glass slides). Moreover, the corresponding pathological reports of the above samples must also be provided. Freshly collected samples, excision, core needle biopsy, resection, incision, punching or forceps biopsies are within the acceptable range (newly-obtained tissues preferred). The aspiration samples (i.e., lack of complete tissue structure and only cell suspension and/or cell smears are provided), brushing samples, cell precipitation samples from pleural or peritoneal effusion are not acceptable. The requirements for tissue samples are provided in laboratory operating manual in detail.

* ECOG performance status score (Appendix II) of 0 or 1 within 7 days before the first dose of invetigational product;
* Life expectancy ≥12 weeks;
* Negative HBsAg; patients with positive HBsAg or HBcAb test results can be enrolled only if Hepatitis B virus (HBV) DNA test results are negative.

  11.Negative HCV antibody; patients with positive HCV antibody or HCV-RNA test results can be enrolled only if ALT and AST are CTCAE v4.03 ≤ grade 1 (i.e., ≤ 3×ULN); subjects concurrently infected with hepatitis B and hepatitis C are excluded.
* Normal function of main organs, and the following criteria are met (within the 14 days before the first injection of investigational product, patients have not received the treatment with blood transfusion, albumin, recombinant human thrombopoietin or colony stimulating factor (CSF)):
* Female subjects must meet the following criteria:

  ① Menopause (defined as no menstruation for at least one year, and no other confirmed reasons other than menopause), or② Received surgical sterilization (ovariectomy and/or hysterectomy), or③ Subjects who are able to bear or father a child must meet the following criteria:
* Serum pregnancy test must be negative within 7 days before the first dosing, and
* Agree to use contraceptive methods with an annual failure rate of < 1% or maintain sexual abstinence (avoid heterosexual intercourse) (from the signing of informed consent form to at least 120 days after the last dose of investigational product) (contraceptive methods with an annual failure rate of < 1% include bilateral tubal ligation, male sterilization, correct use of hormonal contraceptives which may inhibit ovulation, hormone-releasing intrauterine device and copper intrauterine device), and
* Breast-feeding is not allowed.
* Male subjects should meet the criteria below: agree to maintain sexual abstinence (avoid heterosexual intercourse) or use contraceptive methods, with requirements detailed below: if the partners of male subjects have childbearing potential or become pregnant, male subjects must maintain sexual abstinence or use condoms to prevent drug exposure to embryos during administration period of investigational product and within at least 120 days after after the last dose of investigational product. The reliability of sexual abstinence should be evaluated based on the duration of clinical studies, preference of the subjects and daily life style. Regular sexual abstinence (e.g., calendar days, ovulation period, basal body temperature or post-ovulation period contraceptive methods) and coitus interruptus are disqualified contraceptive methods.

Exclusion Criteria:

* Subjects who meet any of the following criteria are not allowed to be enrolled in this study:

  * Subjects who plan to undergo or previously underwent organ or bone marrow transplantation.
  * Uncontrollable pleural effusion, pericardial effusion or ascites after appropriate intervention measures.
  * Subjects with known or screening test-confirmed active central nervous system (CNS) metastasis and/or carcinomatous meningitis; However, the following subjects are allowed to be enrolled: 1. subjects with asymptomatic brain metastasis (i.e. without progressive central nervous system symptoms caused by brain metastatic lesions, without the requirement of corticosteroids treatment, and lesion size ≤1.5cm) are allowed to participate in this study, however, it is necessary to perform regular brain imaging tests for disease sites. 2. subjects with brain metastasis after treatment, and brain metastatic lesions are stable for at least 1 month, without evidence of new or expanded brain metastasis, and steroids are discontinued 3 days prior to the first dose of the investigational product. Stable brain metastasis in this definition should be confirmed before the first dose of the investigational product.
  * Subjects with spinal cord compression which cannot be radically treated through surgery and/or radiotherapy, or subjects previously diagnosed with spinal cord compression with no post-treatment clinical evidence showing stable disease ≥ 1 week before the first dose of the investigational product.
  * Imaging test results show definit tumor invasion of thoracic great vessels.
  * Occurrence of myocardial ischemia above grade Ⅱ , or myocardial infarction, unstable angina pectoris, inadequately controlled arrhythmia (including QTc interval ≥ 450 ms for males, and ≥ 470 ms for females) within half a year before the first dose of the investigational product (QTc interval is calculated based on Fridericia formula).
  * Grade Ⅲ or Ⅳ cardiac dysfunction based on New York Heart Association (NYHA) Functional Classification (appendix Ⅲ) or echocardiography test showing left ventricular ejection fraction (LVEF) < 50%.
  * Presence of peripheral neuropathy with CTCAE v4.03 ≥ grade 2.
  * Infection with human immunodeficiency virus (HIV).
  * Presence of active pulmonary tuberculosis.
  * Previously or currently suffering from interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-related pneumonitis, seriously injured lung function and other conditions which may interfere with the detection and treatment of suspected drug-related pulmonary toxicity.
  * Presence of know active or suspected autoimmune diseases; Patients who have stable status and require no treatment with systemic immunosuppressive therapies are allowed to be enrolled.
  * Treatment with live vaccines within 28 days before the first administration of investigational product.
  * Subjects requiring treatment with systemic corticosteroids (> 10 mg/day prednisone or equivalent dose of similar drugs) or other immunosuppressive therapies within 14 days before the first administration of investigational product or during the study period; However, the following conditions are allowed to be enrolled: in the event of no active autoimmune diseases, inhalation or topical use of steroids or adrenaline alternative treatment of effective dose of prednisone ≤ 10 mg/day are allowed.
  * Presence of any active infection requiring systemic anti-infection treatment within 14 days before the first administration of investigational product.
  * Subjects who have received major surgery within 28 days before the first administration of investigational product, by "major surgery", it meant that the patient needs at least three weeks to recover following the surgery before being able to receive the study treatment. Enrollment through tumor puncture or lymph node biopsy is allowed.
  * Received radical radiotherapy within 3 months before the first administration of investigational product.

Note: palliative radiotherapies for bones or superficial lesions are acceptable. The course of treatment should be in accordance with the local standard and has ended 14 days before the first administration. Radiotherapy covering more than 30% of the bone marrow area is not allowed within 28 days prior to the first dose.

* Other anti-tumor treatments such as chemotherapy, targeted therapy or radiotherapy (excluding palliative radiotherapy) may be received during the study period.
* Previously received treatment with any T cells costimulation or immune checkpoint, including but not limited to cytotoxic T lymphocyte-associated antigen-4 (CTLA-4) inhibitors, PD-1 inhibitors, PD-L1/2 inhibitors or other targeted T cells drugs.
* Subjects are participating in other clinical studies, or the time interval between the initiation of treatment planned in this study and end of investigational product treatment in the previous clinical study is less than 14 days.
* Known serious hypersensitivity history to any monoclonal antibody or the excipients of investigational product.
* Pregnant or lactating women.
* Known history of abuse of psychotropic drugs or drug addiction; Subjects who have stopped drinking are allowed to be enrolled.
* The subjects have other factors which may cause premature termination of this study at the discretion of the investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2019-07-15 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
ORR | up to 2 years
  Objective response rate(assessed by independent radiological review committee (IRRC) based on the RECIST Version 1.1)

SECONDARY OUTCOMES:
ORR | up to 2 years
  Objective response rate (assessed by the investigators based on the RECIST Version 1.1)
ORR | up to 2 years
  Objective response rate (assessed by independent radiological review committee (IRRC) based on the iRECIST)
6-month OS rate | from the date of first dose unitl the date of 6-month
  6-month overall survival rate
OS | from the date of first dose unitl the date of death from any cause，assessed up to 2 years
  Overall survival (OS)
6-month PFS rate | the proportion of subjects who have time interval over 6 months between the first dose and disease progression or death
  6-month progression-free survival (PFS) rate
PFS | from the first dose until firstly confirmed and recorded disease progression or death (whichever occurs earlier),assessed up to 2 years
  Progression-free survival (assessed by independent radiological review committee (IRRC) based on RECIST v1.1, iRECIST)
PFS | from the first dose until firstly confirmed and recorded disease progression or death (whichever occurs earlier),assessed up to 2 years
  Progression-free survival (assessed by the investigators based on RECIST v1.1)
DOR DOR | from the date when CR or PR (whichever recorded earlier) is firstly achieved until the date when disease progression or death is firstly recorded (whichever occurs earlier),assessed up to 2 years
  Duration of response

CONTACTS AND LOCATIONS:
Locations (33):
- China (33):
  - The Second Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Peking University International Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - the 900th Hospital of Joint Logistic Support Force, Fuzhou, Fujian
  - Zhongnan Hospital of Wuhan University, Wuhan, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - First People's Hospital of Fushan, Fushan, Guangdong
  - The First Affiliated Hospital and Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - The First Affiliated Hospital (School of Clinical Medicine), Guangdong Pharmaceutical University, Guangzhou, Guangdong
  - Affiliated Cancer Hospital & Institute, Guangzhou Medical University, Guangzhou, Guangdong
  - the Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Affiliated Hospital of Guangdong Medical University, Zhenjiang, Guangdong
  - Zhongshan city People's Hospital, Zhongshan, Guangdong
  - The Fifth Affiliated Hospital, Sun Yat-sen University, Zhuhai, Guangdong
  - The People's Hospital of Guangxi Zhuangzu Autonomous Region, Nanning, Guangxi
  - Fourth Hospital of Hebei Medical University,, Shijiazhuang, Hebei
  - Harbin Medical University Cancer Hospital,, Harbin, Heilongjiang
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - The Third Xiangya Hospital, Central South University, Changsha, Hunan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Qinhuai Medical District, General Hospital of the eastern theater of the Chinese people's Liberation Army, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - Cancer Hospital of China Medical University, Liaoning Cancer Hospital & Institute, Shenyang, Liaoning
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Shandong Cancer Hospital, Jinan, Shandong
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
  - Sichuan Cancer Hospital & Institute, Sichuan Cancer Center, School of Medicine, University of Electronic Science and Technology of China, Chengdu, Sichuan
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institue and Hospital, Tianjin, Tianjin Municipality
  - Yunnan Cancer Hospital/The Third Affiliated Hospital of Kunming Medical University/Yunnan Cancer Center, Kunming, Yunnan
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Taizhou first people's Hospital, Taizhou, Zhejiang

REFERENCES:
- [Result] Shukui Qin, Jin Li, Haijun Zhong, et al. Efficacy and safety of HLX10, a novel anti-PD-1 antibody, in patients with previously treated unresectable or metastatic microsatellite instability-high or mismatch repair-deficient solid tumors: A single-arm, multicenter, phase 2 study. Journal of Clinical Oncology 2021 39:15_suppl, 2566-2566
- [Result] Qin S, Li J, Zhong H, Jin C, Chen L, Yuan X, Fan Q, Chen K, Cao P, Xiao J, Jiang D, Zhang T, Zhang H, Wang X, Wang W, Han L, Wang Q, Zhu J; Serplulimab-MSI-H Investigators. Serplulimab, a novel anti-PD-1 antibody, in patients with microsatellite instability-high solid tumours: an open-label, single-arm, multicentre, phase II trial. Br J Cancer. 2022 Dec;127(12):2241-2248. doi: 10.1038/s41416-022-02001-3. Epub 2022 Oct 19. PMID 36261583
- See also: Related Info — https://www.nature.com/articles/s41416-022-02001-3